CLINICAL TRIAL: NCT03550430
Title: Study Protocol for a Single-blind Randomized Controlled Trial, Assessing the Specificity of an Alpha/Delta Ratio Neurofeedback Training Protocol in Chronic Tinnitus.
Brief Title: Neurofeedback for Tinnitus - Does Frequency Specificity Matter?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Eriksholm Research Centre (Other); Linkoeping University (Other Government); University Hospital of Gießen and Marburg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neurofeedback for tinnitus
Record Dates: First submitted 2018-05-27; First posted 2018-06-08 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Tinnitus; Subjective Tinnitus; Chronic Tinnitus
Keywords: tinnitus distress; tinnitus intrusiveness; synchronization by loss of inhibition model (SLIM); neurofeedback; alpha/delta neurofeedback; beta/theta neurofeedback; electroencephalography (EEG); tinnitus intensity; tinnitus loudness
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADR neurofeedback (Experimental): Ten ADR neurofeedback training sessions. The first five sessions comprise four training blocks. The latter five sessions consists of five training blocks each. All training blocks are seven minutes in duration. Participants take between two to three sessions each week.
  Interventions: Behavioral: alpha/delta neurofeedback
- BTR neurofeedback (Active Comparator): Ten BTR neurofeedback training sessions. The first five sessions comprise four training blocks. The latter five sessions each consists of five training blocks. All training blocks are seven minutes in duration. Participants take between two to three sessions each week.
  Interventions: Behavioral: beta/theta neurofeedback
- Diary Control Group (Active Comparator): Daily diary completion for two weeks in the period between baseline and end-point assessments (total period baseline to end-point = four weeks).
  Interventions: Other: Diary completion

INTERVENTIONS:
Behavioral: alpha/delta neurofeedback — neurofeedback training protocol seeking to decrease the alpha/delta ratio, by simultaneous rewarding alpha and inhibiting delta activity.
  Arms: ADR neurofeedback
Behavioral: beta/theta neurofeedback — neurofeedback training protocol seeking to decrease the beta/theta ratio, by simultaneous rewarding beta and inhibiting theta activity.
  Arms: BTR neurofeedback
Other: Diary completion — completion of diary relating to participants' experience of tinnitus intensity, interference, coping, harm and disability. Rated three times daily on numerical scale (0 - 10) for two weeks.
  Arms: Diary Control Group

SUMMARY:
This study will evaluate the efficacy of an alpha/delta ratio (ADR) neurofeedback training protocol on tinnitus distress. 1/3 of the participants in the study will undergo ADR neurofeedback training, 1/3 an active comparator, beta/theta ratio (BTR) neurofeedback training, whilst the final 1/3 of participants will fill in daily diaries of tinnitus complaints and symptoms for two weeks.

DETAILED DESCRIPTION:
Tinnitus is hypothesized to originate as a result of a disturbance in the balance of excitatory and inhibitory neurons in central auditory structures. More specifically, inhibitory neurons hyperpolarize, by which their functional role is weakened . Consequently, this allows auditory neurons, deprived of input from a lesioned auditory system, to spontaneously synchronize their activity, resulting in the tinnitus percept.

In the normal functioning auditory system, neurons firing synchronously in the alpha frequency region (8 - 12 Hz) have a gating function of inhibiting task-irrelevant regions in the brain. In people with chronic tinnitus, it has been observed, that alpha activity over temporal regions is weakened, thus leading to the spontaneous activity characterizing the condition. By upregulating alpha activity with neurofeedback training, it is hypothesized that the excitatory/inhibitory balance in temporal regions can be restored, thus minimizing the tinnitus percept.

The coupling or exchange of information of distinct brain regions, leading to an integrated conscious perception, is assumed to be mediated by delta oscillations. In tinnitus, the distress associated with the condition arises as a consequence of coupling prefrontal areas, responsible for allocation of attentional resources with limbic (arousal) and temporal (auditory processing) regions. In neurofeedback, the downregulation of delta activity is hypothesized to lead to a de-coupling of the communication between the areas associated with the distress.

No studies to date have tested the specific role of alpha and delta in the origin and perpetuation of tinnitus distress and intrusiveness. The present study seeks to compensate for this, by comparing an alpha and delta neurofeedback ratio training protocol with one assumed to have no direct association with the pathophysiology of tinnitus.

In addition to the ten neurofeedback training sessions, all participants undergo diagnostic assessments at three time points throughout the trial (pre-neurofeedback training, post-neurofeedback training and at three months follow-up). For the first 40 participants, electroencephalographic (EEG) activity is recorded and cognitive capacity assessed with two attention tests, the Attention Network Test and Sustained Attention Response Task, respectively at all three time points. For the remaining 80 participants, the EEG recording is abandoned, and only cognitive capacity assessed in the pre- post, and follow-up phase of the study.

EEG recording and attention processes is similarly measured in a control group (n=40) at the pre-neurofeedback training stage. The group is comprised of healthy, age and gender matched participants. Their inclusion serve the purpose of comparing the brain activity, both at rest and during cognitive activity between people with- and people without tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Chronic subjective tinnitus, i.e. tinnitus with a duration > 6 months
* At least mild tinnitus distress, corresponding to a score of ≥ 18 on the Tinnitus Handicap Inventory

Exclusion Criteria:

* Moderately severe or severe depression
* Objective tinnitus, where causes are classified according to whether they are vascular or non-vascular in origin
* Current use of psychotropic drugs for a mental health condition
* Bipolar disorder, Attention Deficit Hyperactivity Disorder (ADHD), Psychosis
* Substance abuse
* Current psychotherapeutic treatment for tinnitus, previous biofeedback- or neurofeedback treatment
* A history of seizures, strokes and/or brain hemorrhages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI; Newman, Sandridge, & Jacobson, 1998) | 16 weeks
  Self-report measure of tinnitus handicap assessed pre-intervention, mid-treatment (five sessions), post-intervention and at three month follow-up. The Tinnitus Handicap Inventory is a 25 item questionnaire. Each item is scored 0 - 4 (0 = No, 2 = Sometimes, 4 = Yes), yielding a total between 0 (no handicap) - 100 (catastrophic impact).
Tinnitus Magnitude Index (TMI; Schmidt, Kerns, Griest, Theodoroff, Pietrzak, & Henry, 2014). | 16 weeks
  TMI measures tinnitus intensity, three-item scale assessing self-reported severity, loudness and awareness.
  - Visual analogue scale ranges from 0-10 or 0-100, respectively: item 1 (loudness): Range 0 (not at all strong or loud) to 10 (extremely strong or loud) item 2 (awareness): 0 to 100 in increments of 10, with verbal anchors of 0="never aware" and 100="always aware" item 3 (severity): 0-100 with verbal anchors of 0="no tinnitus present" to 100="the worst tinnitus you can imagine"
  * for all items higher values indicate higher tinnitus magnitude
  * values of the three items can be summed up to a total score. For standardisation, items are converted from 0-100 to 0-10.

SECONDARY OUTCOMES:
Tinnitus Functional Index (TFI; Brüggemann, Szczepek, Kleinjung, Ojo, & Mazurek, 2017) | 16 weeks
  The Tinnitus Functional Index (TFI) is a self-report measure of both perceived severity and negative impact of tinnitus. It covers multiple severity domains including but not exclusively quality of sleep, relaxation, sense of control. The TFI questionnaire consists of 25 items, predominantly scored between 0 - 10 bar item 1 and 3, which are expressed as percentages from 0 - 100%.
Brief Illness Perception Questionnaire (B-IPQ; Broadbent, Petrie, Main, & Weinman, 2006) | 4 weeks
  The B-IPQ is a nine item self-report measure of individual cognitive and emotional representations of illness. It includes the following domains: consequences of the illness; perception of duration of illness; control over illness; treatment control; symptoms; understanding of illness; emotional response and causes.
Insomnia Severity Index (ISI; Bastien, Vallières, & Morin, 2001) | 4 weeks
  A brief scanning measure of insomnia. It consists of 7 items assessing insomnia severity, interference in daily functioning, noticeability of impairment and distress/concern about sleep problems.
Credibility and Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000) | 4 weeks
  a quick and easy-to-administer scale for measuring treatment expectancy and rationale credibility for use in clinical outcome studies
Sustained Attention Response Task (SART; Robertson, Manly, Andrade, Baddeley, & Yiend, 1997) | 16 weeks
  measures the ability to sustain attention
Attention Network Test (ANT; Fan, McCandliss, Sommer, Raz, & Posner, 2002) | 16 weeks
  assesses orienting, alerting and executive attention processing respectively
Patient Health Questionnaire (PHQ-9; Gräfe, Zipfel, Herzog, & Löwe, 2004) | 16 weeks
  Assessment of depressive symptoms

OTHER OUTCOMES:
Satisfaction with treatment | 3 months
  self-developed scale to assess satisfaction with neurofeedback

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Weise, Dr., Principal Investigator — Philipps Universität Marburg
Locations (1):
- Philipps University Marburg, Dept. of Psychology, Division of Clinical Psychology and Psychotherapy, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol
Time Frame: Data available within one year of study completion
Access Criteria: Data access request will be reviewed by the Principal Investigator. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Balkenhol T, Wallhausser-Franke E, Delb W. Psychoacoustic tinnitus loudness and tinnitus-related distress show different associations with oscillatory brain activity. PLoS One. 2013;8(1):e53180. doi: 10.1371/journal.pone.0053180. Epub 2013 Jan 10. PMID 23326394
- [Background] Dohrmann K, Weisz N, Schlee W, Hartmann T, Elbert T. Neurofeedback for treating tinnitus. Prog Brain Res. 2007;166:473-85. doi: 10.1016/S0079-6123(07)66046-4. PMID 17956812
- [Background] Weisz N, Dohrmann K, Elbert T. The relevance of spontaneous activity for the coding of the tinnitus sensation. Prog Brain Res. 2007;166:61-70. doi: 10.1016/S0079-6123(07)66006-3. PMID 17956772
- [Background] Weisz N, Hartmann T, Muller N, Lorenz I, Obleser J. Alpha rhythms in audition: cognitive and clinical perspectives. Front Psychol. 2011 Apr 26;2:73. doi: 10.3389/fpsyg.2011.00073. eCollection 2011. PMID 21687444
- [Background] Newman CW, Sandridge SA, Jacobson GP. Psychometric adequacy of the Tinnitus Handicap Inventory (THI) for evaluating treatment outcome. J Am Acad Audiol. 1998 Apr;9(2):153-60. PMID 9564679
- [Background] Schmidt CJ, Kerns RD, Griest S, Theodoroff SM, Pietrzak RH, Henry JA. Toward development of a tinnitus magnitude index. Ear Hear. 2014 Jul-Aug;35(4):476-84. doi: 10.1097/AUD.0000000000000017. PMID 24603542
- [Background] Bruggemann P, Szczepek AJ, Kleinjung T, Ojo M, Mazurek B. [Validation of the German Version of Tinnitus Functional Index (TFI)]. Laryngorhinootologie. 2017 Sep;96(9):615-619. doi: 10.1055/s-0042-122342. Epub 2017 May 12. German. PMID 28499301
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. J Cogn Neurosci. 2002 Apr 1;14(3):340-7. doi: 10.1162/089892902317361886. PMID 11970796
- [Background] Robertson IH, Manly T, Andrade J, Baddeley BT, Yiend J. 'Oops!': performance correlates of everyday attentional failures in traumatic brain injured and normal subjects. Neuropsychologia. 1997 Jun;35(6):747-58. doi: 10.1016/s0028-3932(97)00015-8. PMID 9204482
- [Background] Gräfe, K., Zipfel, S., Herzog, W., & Löwe, B. (2004). Screening psychischer Störungen mit dem "Gesundheitsfragebogen für Patienten (PHQ-D)". Diagnostica, 50(4), 171-181.
- [Derived] Jensen M, Huttenrauch E, Schmidt J, Andersson G, Chavanon ML, Weise C. Neurofeedback for tinnitus: study protocol for a randomised controlled trial assessing the specificity of an alpha/delta neurofeedback training protocol in alleviating both sound perception and psychological distress in a cohort of chronic tinnitus sufferers. Trials. 2020 May 5;21(1):382. doi: 10.1186/s13063-020-04309-y. PMID 32370767